CLINICAL TRIAL: NCT01111032
Title: Comparison of Two-treadmill Test Protocols to Evaluate Endurance in People With Cancer.
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Oren Cheifetz, Clinical Specialist - Physiotherapy, McMaster University
Organization: McMaster University (Other)
Other Study IDs: Treadmill Comparison
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Cancer
Keywords: Treadmill; Exercise; Cancer; Validity; Reliability
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treadmill test

SUMMARY:
During this study the investigators will compare the use of two treadmill tests in people diagnosed with cancer. The STEEP treadmill protocol is often used to evaluate the endurance of people diagnosed with cancer, however, since it is based on step increases in speed or ramp, it may not related to normal function. The new test, which is based on the body response to increased activity has not been used with people with cancer but may provide a better approximation of endurance demands during daily function. Our question is whether the new treadmill test can be used to evaluate aerobic function with people with cancer better than the STEEP treadmill test.

ELIGIBILITY:
Inclusion Criteria:

* Participants are required to be adults (age 16 or over),
* Diagnosed with cancer, at any stage of treatment (during or after treatment),
* Able to follow instructions in English, and provide informed consent.
* Participants need to be considered "well" to participate. A "well participant" has been defined as a cancer survivor who is living at home, able to ambulate independently without a gait aid (single point cane is acceptable), has no acute medical conditions, and passes pre-exercise safety screening.

Exclusion Criteria:

* Cancer survivors with metastatic disease.
* Cancer survivors who are defined as unwell.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult well cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
STEEP treadmill test | 1 hour
  Treadmill test for endurance. Lasts approx 15 min with 45 min recovery

CONTACTS AND LOCATIONS:
Overall Officials: Oren Cheifetz, M.Sc. PT, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Henderson Campus, Hamilton, Ontario, Canada